CLINICAL TRIAL: NCT01832935
Title: Cost Effectiveness of Glargine Insulin Versus NPH Insulin in Diabetic Patients in Iran
Brief Title: Cost Effectiveness of Glargine Insulin Versus NPH Insulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Esteghamati, professor alireza esteghamati, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 89-123
Record Dates: First submitted 2013-04-11; First posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Glargin; NPH; Cost-effectiveness
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin, Isophane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- insulin glargine (Active Comparator): patients receiving variable doses of Insulin glargine.start with 0.2 to 0.6unit per kg
  Interventions: Drug: insulin glargine
- Insulin NPH (Active Comparator): patients receiving Variable doses Of Insulin NPH Start with 0.2 to 0.6 unit per kg
  Interventions: Drug: Insulin NPH

INTERVENTIONS:
Drug: insulin glargine — The starting dose of insulin Glargine was 24 units per day (0.2-0.6 unit/kg) in 2 divided doses
  Other Names: Lantus
  Arms: insulin glargine
Drug: Insulin NPH — The starting dose of insulin NPH was 24 units per day (0.2-0.6 unit/kg) in 2 divided doses
  Arms: Insulin NPH

SUMMARY:
Glycemic control is fundamental in the management of diabetes mellitus .If lifestyle intervention and full tolerated doses of one or two oral glucose lowering drugs (OGLDs) fail to achieve or sustain glycemic goals, insulin should be initiated. New insulin analogs are generated to improve glycemic control .New insulin analogs are generated to improve glycemic control,However, the cost of these analogs is a major problem .The aim of this piggy back evaluation was to assess the effect of Glargine insuline versus NPH plus regular human insulin on metabolic control as well as its cost-effectiveness in people with type 2 diabetes in the Iranian setting.

DETAILED DESCRIPTION:
This was a randomized double blind controlled clinical trial of 12months on subjects with type 2 diabetes. Two hundred diabetic subjects, 18-65 years of age, were included in the study. Subjects were willing to initiate insulin therapy and had A1C >8.0%. Any current and prior medications were acceptable for participant inclusion other than any type of insulin being evaluated. Demographic and anthropometric variables were recorded. Paraclinical data including glucose and lipid profile were measured every three months.In addition, quality of life was assessed with self-administered standard EQ-5D questionnaire.

Subjects were excluded for any of the following criteria: Alteration in insulin sensitivity such as major surgery, infection, renal failure (Glomerular Filtration Rate < 50), glucocorticoid treatment, recent (within 2 weeks) serious hypoglycemic episode (requires assistance of another), simultaneous participating in another clinical study, using any type of insulin, sight or hearing impaired, active proliferative retinopathy or maculopathy require treatment within 6 months prior to screening, breast feeding, pregnancy or nursing of the intention of becoming pregnant or not using adequate contraceptive measures.

Participants were recruited between July 2011 and October 2012. They were randomly allocated to two groups using a simple randomization method The insulin therapies were prescribed by a physician in the clinic. The starting dose of insulin Glargine was 24 units per day (0.2-0.6 unit/kg) in 2 divided doses in the intervention group. The control group received NPH/Reg insulin (2:1) with initiation dose of 0.2-0.6 unit/kg in 2 divided doses.Two-thirds of the dose was given before breakfast and the remainder before dinner. In the study, insulin analogues were used in accordance with the licensed approval from the local regulatory authority. Changes to OGLDs at the time of starting the insulin analogue, or thereafter, were entirely at the discretion of the participant and physician. Paraclinical data were measured in a referral laboratory every three months. Trial visits were defined as 0, 12, 24, 36 and 48 weeks from baseline. All participants were asked to record their 7-point blood glucose values in three consecutive days before each visit. Seven-point self-monitoring blood glucose includes three pre-meals, three post-meals, and bedtime blood glucose values during each day.Insulin doses were adjusted by a titration regimen according to self-monitored blood glucose.For both groups, treatment goals were as follows: fasting blood glucose of 80-120 mg/dl, postprandial glucose <160 mg/dl, A1C<7% We collected medical costs of each patient by a checklist. All patients had been asked to attend in our clinic every one month during the study. Clinical events or hospital episodes and also all related costs were determined at each visit. Any pharmaceutical, laboratory/diagnostic and rehabilitative care, as well as any contact with specialists, general practitioners, nurses, opticians, podiatrists, and dieticians were recorded for patients with/without complication.Finally total costs were calculated.

Direct nonmedical costs:

Any services such as transportation for patients and their family to clinic and taking care of dependents were assessed for non-medical expenditures by a patient self-estimate questionnaire.

Indirect costs:

The lost productivity costs due to health problems of diabetes were determined by days absent from work, poor work performance, low earnings capacity from disabilities, and mortality. We calculated number of days in each visit who could not be present in their job because of diabetes related health care. The average net hourly wage was asked from each patient. For unemployed patients, we considered average wage of population who were economically active and in employment. Lost earnings owing to premature mortality were defined as the mortality costs. Costs from health provider perspective, were converted from Iranian Rials (IRR) into USA dollar (USD) at an official exchange rate of 12,260 IRR/1USD 2012 to have an international comparison (Central Bank of Iran).

ELIGIBILITY:
Inclusion Criteria:

* diabetes type 2
* HbA1c 8% or higher
* age 18 to 65

Exclusion Criteria:

* alteration in insulin sensitivity such as major surgery, infection, renal failure (Glomerular Filtration Rate < 50),
* glucocorticoid treatment,
* recent (within 2 weeks) serious hypoglycemic episode (requires assistance of another),
* simultaneous participating in another clinical study,
* using any type of insulin,
* sight or hearing impaired,
* active proliferative retinopathy or maculopathy require treatment within 6 months prior to screening,
* breast feeding,
* pregnancy or nursing of the intention of becoming pregnant or
* not using adequate contraceptive measures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number Of Hypoglycemic events | 3 months
  The Number Of Hypoglycemic Events That Happend For Patients During Taking Both Insulines

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Esteghamati, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Tehran, Tehran Province, Iran